CLINICAL TRIAL: NCT03522298
Title: A Phase 2 Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of the PI3K/mTOR Inhibitor Paxalisib (GDC-0084) Administered to Patients With Glioblastoma Characterized by Unmethylated O6-methylguanine-methyltransferase Promoter Status Following Surgical Resection and Standard Concomitant Chemoradiation Therapy With Temozolomide
Brief Title: Safety, Pharmacokinetics and Efficacy of Paxalisib (GDC-0084) in Newly-diagnosed Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kazia Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVGN-0084-201
Record Dates: First submitted 2018-03-20; First posted 2018-05-11 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma, Adult
Keywords: newly diagnosed; unmethylated O6 methylguanine-methyltransferase (MGMT) promoter status
MeSH Terms: conditions — Glioblastoma | interventions — GDC-0084

STUDY DESIGN:
Intervention Model Description: This phase 2 study comprises an open-label, multicenter, dose-escalation and expansion study to assess the safety, tolerability, RP2D, PK and clinical activity of paxalisib in patients with newly-diagnosed GBM with unmethylated MGMT promoter status as adjuvant therapy following surgical resection and initial chemoradiation with TMZ.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion Cohorts (Experimental): This is an open-label study.
  Patients in Stage 1 will be enrolled and sequentially assigned to a dose cohort.
  The initial cohort will receive an oral dose of 60 mg paxalisib QD (4 x 15 mg capsules). Patients of future dose cohorts will receive paxalisib at increasing levels with 15 mg steps until a dose-limiting toxicity occurs (DLT) occurs. The dose level where <1/3 of the patients exhibit a DLT will be determined the Maximum Tolerated Dose (MTD).
  In stage 1, dose escalation will occur for QD dosing.
  In stage 2, the expansion phase, patients will receive doses of oral paxalisib at the MTD in stage 1, until disease progression or an unacceptable toxicity, whichever occurs first.
  Patients will be randomized in a 1:1 ratio to fed or fasted schedules.
  Interventions: Drug: Paxalisib (GDC-0084)

INTERVENTIONS:
Drug: Paxalisib (GDC-0084) — Patients will be dosed orally with paxalisib (GDC-0084) capsules (15-mg each) at the dose and schedule to which they are assigned.

SUMMARY:
This protocol has a 2-part design:

This phase 2 study is an open-label, multicenter, dose-escalation and expansion study to assess the safety, tolerability, recommended phase 2 dose (RP2D), pharmacokinetics (PK) and clinical activity of paxalisib in patients with newly-diagnosed glioblastoma (GBM) with unmethylated MGMT promoter status as adjuvant therapy following surgical resection and initial chemoradiation with temozolomide (TMZ).

DETAILED DESCRIPTION:
Stage 1 Dose-Escalation and Maximum Tolerated Dose The dose-escalation portion of the study (Stage 1) will use a standard "3 + 3" design to determine the MTD for QD dosing.

Approximately 6 - 12 patients with newly diagnosed GBM will be enrolled in Stage 1.

The MTD for QD dosing will be determined. The initial dose level for QD dosing will be 60 mg (Dose Level 0). This dose is based on the phase 1 findings outlined in the rationale in the protocol, adding 1 dose level to test for a potential MTD increase.

Dose-escalation will occur in Stage 1:

* The initial dose (Dose Level 0) for QD MTD determination in Step 1 will be 60 mg. Dose levels will increase in 15 mg steps;
* The dose-escalation portion of the study (Stage 1) will use a standard "3 + 3" design to assess the safety, tolerability, and PK of paxalisib administered orally in 28-day cycles;

Decisions regarding dose-escalation and selection will be made by a Cohort Review Committee (CRC).

All AEs, including DLTs, will be reported, with severity assessed according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03.

After determination of the MTD, patients continue to receive their protocol-assigned dose levels of paxalisib until progression of their disease or an unacceptable toxicity, whichever occurs first.

Stage 2 Expansion stage (2) of the study will be a two-arm, randomized, open-label expansion study to further characterize the safety, tolerability and PK of paxalisib as well as to provide a preliminary assessment of single-agent activity of paxalisib in patients with GBM. Approximately 20 patients will be enrolled in the expansion cohort in 2 treatment arms (10 per am) to examine the PK of paxalisib in fed and fasted-conditions, according to the defined study eligibility criteria.

Stage 2 of the study will be initiated with recruitment of new patients as soon as the MTD has been determined.

Patients enrolled in Stage 2 may continue the study at the dose allocated until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following inclusion criteria to be eligible for enrollment into the study:

1. Age ≥ 18 years;
2. Life expectancy > 12 weeks;
3. Present with histologically confirmed intracranial (supratentorial) unmethylated MGMT promotor status GBM (WHO Grade lV astrocytoma) with a MGMT status that has been confirmed by validated PCR or validated alternate genomic analysis;
4. Have undergone maximal surgical resection of their tumor and within 6 weeks of surgery received initial treatment with XRT/TMZ which consisted of XRT by external beam to a partial brain field in daily fractions of 2.0 Gray (Gy), to a planned total dose to the tumor of 60.0 Gy, in conjunction with TMZ oral QD 75 mg/m2 in accordance with the Stupp regimen;
5. Must have measurable disease, according to RANO criteria for inclusion in the expansion cohort. Patients with non-measurable disease can be included in the dose-escalation cohorts;
6. KPS ≥ 70;
7. Cranial magnetic resonance imaging (MRI) must have been performed within 7 days prior to or on the day of the Randomization/Week 1 Visit;
8. Stable or decreasing corticosteroid dose within 7 days prior to the first dose;
9. Adequate bone marrow/hematological function within 7 days prior to Day 1;
10. Adequate liver and renal function within 14 days prior to Day 1;
11. International normalized ratio (INR) or prothrombin time (PT) (secs) and activated partial thromboplastin time (aPTT) within 7 days prior to randomization:
12. Patients must be willing to forego other drug therapy against the tumor while enrolled in the study.

Exclusion Criteria:

1. Previous radiotherapy to the brain or cytotoxic drug therapy (including Gliadel® wafers) in addition to the required postoperative radiation plus TMZ, non-cytotoxic drug therapy, or experimental drug therapy directed against the brain tumor prior to this regimen, will be excluded. Patients may have received or be receiving corticosteroids, analgesics, and other drugs to treat symptoms or prevent complications but the dose must be stable at treatment start. NOTE: 5 aminolevulinic acid-mediated photodynamic therapy administered prior to surgery to aid in optimal surgical resection is not considered a chemotherapy agent;
2. Any prior or anticipated concomitant treatment involving a medical device (such as Optune®) applying tumor treating fields (TTF);
3. QT interval time of ≥ 470 msec;
4. Undetermined/indeterminate MGMT status;
5. Diabetic patients; prediabetic patients treated with metformin;
6. Use of any CYP3A4 inducing or inhibiting agents;
7. Significant medical illnesses;
8. Women who are pregnant or who are lactating;
9. Diagnosed with infratentorial GBM, a tumor outside of brain or gliomatosis cerebri;
10. Evidence of recent hemorrhage on postoperative MRI of the brain;
11. Any previous malignancy; except for adequately controlled limited basal cell carcinoma of the skin, squamous carcinoma of the skin or carcinoma in situ of the cervix, or one which has been absent for ≥3 years;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Garner, MD, Study Director — Kazia Therapeutics Limited
Locations (6):
- United States (6):
  - University of California Los Angeles - Jonsson Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - University of Oklahoma Health Sciences Center (Stephenson Cancer Center), Oklahoma City, Oklahoma
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, multicenter dose-escalation study with expansion. This study comprised 2 stages, Stage 1 (dose escalation) and Stage 2 (dose expansion and fed/fasted investigation)
Pre-assignment Details: Each stage started with a screening period (Days -28 to -1), followed by treatment and follow-up periods
Groups:
- Dose-escalating Cohort 1: Paxalisib 60mg: Stage 1, Cohort 1
  Participants were administered 60 mg paxalisib (4 ×15 mg capsules) orally once per day in 28-day cycles. Participants fasted for 10 hours pre-dose and for 4 hours post-dose on days when they underwent PK assessments (Cycle 1 Day 1 and Cycle 2 Day 1). On all other days doses were administered at least 1 hour before or 2 hours after food to ensure the study medication was taken on an empty stomach
- Dose-escalating Cohort 2: Paxalisib 75 mg: Participants were administered 75 mg paxalisib (5 ×15 mg capsules) orally once per day in 28-day cycles. Participants fasted for 10 hours pre-dose and for 4 hours post-dose on days when they underwent PK assessments (Cycle 1 Day 1 and Cycle 2 Day 1). On all other days doses were administered at least 1 hour before or 2 hours after food to ensure the study medication was taken on an empty stomach.
- Expansion Cohort: Paxalisib 60mg (Fed): Participants were administered 60 mg paxalisib (4 ×15 mg capsules) orally once per day in 28-day cycles. Participants consumed a high-fat, high-calorie meal approximately 30 minutes prior to dosing, and fasted thereafter for at least 4 hours on days when they underwent PK assessments (Cycle 1 Day 1 and Cycle 2 Day 1). On all other days doses were administered at least 1 hour before or 2 hours after food to ensure the study medication was taken on an empty stomach.
- Expansion Cohort: Paxalisib 60mg (Fasted): Stage 2, Fasted
  Participants were administered 60 mg paxalisib (4 ×15 mg capsules) orally once per day in 28-day cycles. Participants fasted for 10 hours pre-dose and for 4 hours post-dose on days when they underwent PK assessments (Cycle 1 Day 1 and Cycle 2 Day 1). On all other days doses were administered at least 1 hour before or 2 hours after food to ensure the study medication was taken on an empty stomach.
Period: Overall Study
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Started | 3 | 6 | 10 | 11
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 10 | 11
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Death | 2 | 4 | 8 | 8
Not completed — Patient decision | 0 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: ITT population The intent-to-treat (ITT) population consisted of all patients who were enrolled in the study, whether in Stage 1 or Stage 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted) | Total
Number analyzed (Participants) | 3 | 6 | 10 | 11 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (15.72) | 56 (9.30) | 56 (12.51) | 59.5 (9.46) | 58.5 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 4 | 9
  Male | 3 | 4 | 7 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 3 | 5 | 10 | 10 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 4 | 9 | 10 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 10 | 11 | 30
Time since diagnosis [Mean (Standard Deviation); unit: months] | 3.68 (0.553) | 4.33 (1.137) | 3.64 (0.358) | 3.56 (0.318) | 3.75 (0.637)
Type of surgery [Count of Participants; unit: Participants]
  Biopsy (Patients later had a complete resection) | 0 | 0 | 1 | 1 | 2
  Complete resection | 2 | 4 | 9 | 7 | 22
  Partial resection | 1 | 2 | 0 | 2 | 5
  Other (stereotactic biopsy) | 0 | 0 | 0 | 1 | 1
Histological diagnosis [Count of Participants; unit: Participants] | 3 | 6 | 10 | 11 | 30
Karnofsky Performance Status [Count of Participants; unit: Participants] — 100: Normal no complaints; no evidence of disease 90: Able to carry on normal activity; minor signs or symptoms of disease 80: Normal activity with effort; some signs or symptoms of disease 70: Cares for self; unable to carry on normal activity or to do active work 60: Requires occasional assistance, but is able to care for most of his personal needs 50: Requires considerable assistance and frequent medical care 40 or less: Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly.
  Participants
    100 | 0 | 0 | 2 | 0 | 2
    90 | 0 | 5 | 4 | 10 | 19
    80 | 3 | 0 | 2 | 0 | 5
    70 | 0 | 1 | 2 | 1 | 4
    60 | 0 | 0 | 0 | 0 | 0
    50 | 0 | 0 | 0 | 0 | 0
    40 or less | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as a Grade 3 or 4 toxicity occurring within the DLT assessment window and assessed to be probably or possibly related to paxalisib. DLTs were graded using the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. CTCAE Grade 3 is a severe adverse event (AE) and Grade 4 is a life-threatening or disabling AE. DLTs were collected to determine the maximum tolerated dose (MTD), which was defined as the dose level below the dose at which less than 33% of participants experienced a DLT.
Time Frame: Cycle 1, Days 1-28
Population: All participants in Stage 1 (dose-escalating cohorts 1 and 2) who received at least one dose of paxalisib
Measure: Count of Participants; unit: Participants
Groups:
- Dose-escalating Cohort 2: Paxalisib 75 mg: Stage 1, Cohort 2
  Participants were administered 75 mg paxalisib (5 ×15 mg capsules) orally once per day in 28-day cycles. Participants fasted for 10 hours pre-dose and for 4 hours post-dose on days when they underwent PK assessments (Cycle 1 Day 1 and Cycle 2 Day 1). On all other days doses were administered at least 1 hour before or 2 hours after food to ensure the study medication was taken on an empty stomach.
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg
Number analyzed (Participants) | 3 | 6
Participants | 0 | 2

2. Secondary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs)
Description: The toxicity assessments were made according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. A TEAE is any AE occurring or worsening on/after the first study drug dose and within 28 days after the last dose date. The number of participants with Grade 1 to 5 TEAEs are reported here. Specific Adverse Event terms are provided in the Adverse Event module
Time Frame: 24 months
Population: Safety population: All participants who received at least 1 dose of paxalisib
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
Participants | 3 | 6 | 10 | 11

3. Secondary Outcome: Incidence of Serious Adverse Events (SAEs)
Description: An SAE is any AE that meets one or more of the following: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; requires intervention to prevent permanent impairment or damage. Specific AE terms are provided in the Adverse Event module
Time Frame: 24 months
Population: Safety population: All participants who received at least 1 dose of paxalisib
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
Participants | 2 | 5 | 6 | 5

4. Secondary Outcome: Incidence of Treatment-emergent Grade 3/4 Treatment Emergent Adverse Events
Description: Treatment emergent Adverse Events were graded using the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. CTCAE Grade 3 is a severe adverse event (AE) and Grade 4 is a life-threatening or disabling AE. Participants are counted at the highest grade TEAE that they experienced.
Time Frame: 24 months
Population: Safety population: All participants who received at least 1 dose of paxalisib
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
Participants
  Grade 1 or 2 | 0 | 0 | 1 | 0
  Grade 3 | 3 | 3 | 9 | 10
  Grade 4 | 0 | 3 | 0 | 1

5. Secondary Outcome: Number of Participants Who Experienced a Change in Electrocardiogram (ECG) Parameter QTc
Description: A change in ECG parameter QTc was defined as an increase of QTc to a value ≥ 500 msec or a change from baseline of at least 60 msec.
Time Frame: 24 months
Population: Safety population: All participants who received at least 1 dose of paxalisib
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Who Experienced a Change Left Ventricular Ejection Fraction
Description: A change in left ventricular ejection fraction (LVEF) was defined as a reduction in LVEF to a value of ≤ 45% from baseline.
Time Frame: 24 months
Population: Safety population: All participants who received at least 1 dose of paxalisib
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
Participants | 0 | 0 | 0 | 1

7. Secondary Outcome: Progression-free Survival Interval Using Using mRANO Criteria/Investigator Review.
Description: Progression-free survival is defined as the duration of time from start of treatment to time of progression or death, whichever comes first.
Time Frame: 24 months
Population: Intention to treat: All patients who were enrolled in the study, whether in Stage 1 or Stage 2.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
Months | 14.5 [3.3 to 25.7] | 4.7 [1.8 to 27.4] | 7.0 [1.0 to 13.2] | 5.5 [2.0 to 11.8]

8. Secondary Outcome: Overall Survival Using RANO Criteria.
Description: Overall survival is defined as the duration of time from the first day of study treatment until the date of death.
Time Frame: 24 months
Population: Intention to treat: All patients who were enrolled in the study, whether in Stage 1 or Stage 2.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
Months | 20.1 [14.4 to 25.7] | 11.8 [4.4 to 37.5] | 12.0 [7.6 to 17.6] | 9.8 [2.0 to 15.1]

9. Other Pre Specified Outcome: Pharmacokinetics of Paxalisib as Area Under the Curve From Time 0 to Last Measurable Time Point (AUC0-last) and/or Area Under the Curve From Time 0 to Infinity (AUC0-inf).
Description: Blood samples were obtained and plasma concentrations were determined using a validated high-pressure liquid chromatography method. Samples were obtained: prior to the initial dose on Cycle 1 Day 1 and then at 30 minutes, and at 1, 2, 3, 4, 6 8 and 24 hours post dose.
Time Frame: 24 hours
Population: Safety population: All participants who received at least 1 dose of paxalisib
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*h
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
ng/mL*h | 1180 (36.6) | 1120 (91.4) | 2190 (34.5) | 1640 (67.1)

10. Other Pre Specified Outcome: Maximum Observed Plasma Concentration of Paxalisib (Cmax)
Description: as for outcome 9
Time Frame: 24 hours
Population: Safety population: All participants who received at least 1 dose of paxalisib
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
ng/mL | 174 (108) | 118 (67.4) | 176 (24.2) | 114 (44.2)

11. Other Pre Specified Outcome: Pharmacokinetics of Paxalisib as Time to Reach Cmax (Tmax).
Description: as for outcome 9
Time Frame: 24 hours
Population: Safety population: All participants who received at least 1 dose of paxalisib
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
Hours | 3.00 [2.00 to 5.42] | 2.50 [1.95 to 4.00] | 4.00 [2.80 to 8.00] | 3.93 [3.00 to 8.00]

12. Other Pre Specified Outcome: Change in FDG-PET Uptake in Response to Paxalisib in Patients With Measurable Disease.
Description: FDG-PET imaging was obtained using a stand-alone PET or combined PET/computed tomography (CT) scanner, or hybrid PET/MRI systems and the and mean FDG-PET standard uptake value quantified
Time Frame: Cycle 1, Day 3
Population: All participants in Stage 2 (dose-expansion cohorts) who received at least one dose of paxalisib and had measurable disease
Measure: Mean (Standard Deviation); unit: standardized uptake value
Groups:
- Expansion Cohort: Paxalisib 60mg (Fed): Stage 2, Fed
  Participants were administered 60 mg paxalisib (4 ×15 mg capsules) orally once per day in 28-day cycles. Participants consumed a high-fat, high-calorie meal approximately 30 minutes prior to dosing, and fasted thereafter for at least 4 hours on days when they underwent PK assessments (Cycle 1 Day 1 and Cycle 2 Day 1). On all other days doses were administered at least 1 hour before or 2 hours after food to ensure the study medication was taken on an empty stomach.
Arm/Group | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 5 | 5
standardized uptake value | 0.036 (0.7523) | -0.442 (0.3517)

13. Other Pre Specified Outcome: Change in FDG-PET Uptake in Response to Paxalisib in Patients With Measurable Disease
Description: as for outcome 12
Time Frame: Cycle 1, Day 7
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: standardized uptake value
Arm/Group | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 5 | 5
standardized uptake value | -0.366 (1.1814) | -0.432 (0.5963)

14. Other Pre Specified Outcome: Disease Control Rate.
Description: Response to treatment was assessed by MRI using the response assessment in neuro-oncology (RANO) criteria based on the assessment of the MRI scan and clinical features. The DCR is defined as the proportion of patients achieving a confirmed best overall response of complete response (CR; disappearance of all enhancing disease, clinically stable/improved), partial response (PR; 50% or more decrease in measurable enhancing lesions, clinically stable/improved), or stable disease (SD, does not qualify for CR or PR, does not qualify for disease progression, clinically stable). To be assigned a status of CR, PR or SD patients need to have two consecutive assessments of CR, PR or SD. To be assigned a best overall response of SD patients must have a minimum duration of SD of at least 6 weeks.
Time Frame: 24 months
Population: Safety population: All participants who received at least 1 dose of paxalisib
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
Number analyzed (Participants) | 3 | 6 | 10 | 11
Participants | 3 | 4 | 8 | 9

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events may have been volunteered spontaneously by the patient, discovered as a result of general questioning by the study staff, or determined by physical examination. Adverse events were followed until they resolved, were stable, or until the patient's last study visit or were lost to follow-up.
Arm/Group | Dose-escalating Cohort 1: Paxalisib 60mg | Dose-escalating Cohort 2: Paxalisib 75 mg | Expansion Cohort: Paxalisib 60mg (Fed) | Expansion Cohort: Paxalisib 60mg (Fasted)
All-Cause Mortality (participants affected / at risk) | 2/3 | 4/6 | 8/10 | 8/11
Serious Adverse Events (participants affected / at risk) | 2/3 | 5/6 | 6/10 | 5/11
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 10/10 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-escalating Cohort 1: Paxalisib 60mg (N=3) | Dose-escalating Cohort 2: Paxalisib 75 mg (N=6) | Expansion Cohort: Paxalisib 60mg (Fed) (N=10) | Expansion Cohort: Paxalisib 60mg (Fasted) (N=11)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central nervous system haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reversible cerebral vasoconstriction syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-escalating Cohort 1: Paxalisib 60mg (N=3) | Dose-escalating Cohort 2: Paxalisib 75 mg (N=6) | Expansion Cohort: Paxalisib 60mg (Fed) (N=10) | Expansion Cohort: Paxalisib 60mg (Fasted) (N=11)
Fatigue (General disorders) | 3 (7) | 4 (8) | 6 (10) | 9 (13)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 2 (4) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (8) | 6 (10) | 4 (5)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (3) | 4 (4) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (7) | 2 (2) | 5 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 5 (7) | 6 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (3) | 5 (10) | 3 (4) | 4 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 4 (4) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 1 (1) | 1 (2)
Hypertrigliceridaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (3) | 2 (2) | 5 (8)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5) | 2 (3) | 4 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 2 (3) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (4) | 0 (0) | 1 (4) | 2 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (2)
Cognitive disorder (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 4 (4) | 2 (2) | 1 (3)
Neutrophil count decreased (Investigations) | 1 (3) | 2 (6) | 2 (3) | 3 (5)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 3 (12) | 1 (3) | 1 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 1 (2) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 2 (2) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 2 (2) | 0 (0) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/98/NCT03522298/Prot_SAP_000.pdf